CLINICAL TRIAL: NCT07271394
Title: The Impact of Methylprednisolone Sodium Succinate on Postoperative Delirium in Elderly Patients Undergoing Abdominal Surgery: A Target Trial Emulation Study
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jingsheng Lou, Professor, Chinese PLA General Hospital
Other Study IDs: YXM02
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Delirium (POD)
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged ≥ 65 years undergoing abdominal surgery
  Interventions: Drug: Administration of methylprednisolone sodium succinate during general anesthesia induction; Drug: No administration of methylprednisolone sodium succinate during general anesthesia induction

INTERVENTIONS:
Drug: Administration of methylprednisolone sodium succinate during general anesthesia induction — Administration of methylprednisolone sodium succinate during general anesthesia induction
Drug: No administration of methylprednisolone sodium succinate during general anesthesia induction — No administration of methylprednisolone sodium succinate during general anesthesia induction

SUMMARY:
Glucocorticoids can be used to inhibit postoperative systemic inflammatory response syndrome. They may reduce the risk of major complications and mortality. Previous studies on the effect of glucocorticoids on postoperative cognitive dysfunction may lack generalizability due to short follow-up periods for cognitive function after surgery, insufficient follow-up results of cognitive function throughout the entire hospitalization, and a single surgical approach. Clinical evidence provided by previous randomized controlled trials may be biased due to loss-to-follow-up rates caused by researchers' failure to timely follow up on cognitive dysfunction outcomes. Most previous randomized controlled trials investigating the effect of glucocorticoids on postoperative delirium have limitations, mainly including small sample sizes and limited statistical power. Given the high cost of conducting large-scale randomized controlled trials involving various types of perioperative abdominal surgeries in elderly patients and the practical difficulty of reducing loss-to-follow-up rates, there is an urgent need to find alternative approaches. In this study, we extracted data from the in-hospital electronic medical record system and conducted a target simulation trial based on the designed randomized controlled trial protocol investigating the effect of methylprednisolone sodium succinate on postoperative delirium in elderly patients undergoing abdominal surgery. Using existing data, we analyzed whether administration of methylprednisolone sodium succinate during anesthesia induction has an impact on the incidence of postoperative delirium in elderly patients undergoing abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1、Age ≥ 65 years; 2、Patients undergoing abdominal surgery under general anesthesia, including gynecological, hepatobiliary, gastrointestinal, and urological surgeries.

Exclusion Criteria:

* 1、Patients with American Society of Anesthesiologists (ASA) physical status classification ≥ Ⅳ (including Class Ⅳ);2、Patients admitted to the intensive care unit (ICU) postoperatively; 3、Patients with a preoperative history of schizophrenia, epilepsy, or Parkinson's disease;4、Patients with diseases requiring hormone therapy for more than 7 days within 1 year prior to surgery; 5、Patients unable to communicate preoperatively (due to coma, severe dementia, or language/hearing impairment) and those with a Mini-Mental State Examination (MMSE) score < 26;6、Patients with any cerebrovascular event within the past 3 years; 7、Patients who underwent general anesthesia surgery within the past 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥ 65 years undergoing abdominal surgery
Sampling Method: Probability Sample
Enrollment: 25800 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium within 3 days postoperatively | within 3 days postoperatively

SECONDARY OUTCOMES:
Incidence of postoperative delirium within 7 days postoperatively | within 7 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China